CLINICAL TRIAL: NCT06106932
Title: The Effects of GnRH-a on Angiogenesis of Endometriosis
Brief Title: GnRH-a on Angiogenesis of Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Apostolos Kaponis, Associate Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-05-2015/83
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Angiogenesis; Endometriosis
Keywords: Endometriosis; Angiogenesis; GnRH-a; VEGF; SP1
MeSH Terms: conditions — Endometriosis | interventions — Leuprolide

STUDY DESIGN:
Intervention Model Description: This was a prospective randomized follow up study with analysis of ovarian samples derived from GnRH agonists-treated and non-treated women before surgery. The randomization was performed by accessing a central internet-based randomization program. The random allocation sequence and the assignment of the participants to interventions were made by 2 of the authors [A.K. and S.K].
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH-a + (Active Comparator): Group A [GnRHa+] consisted of 30 women with a mean age of 35.5 years and a mean BMI of 27 kg/m2. Seventeen of them were stage 2 and 13 were stage 3 endometriosis. They received GnRH-a [leuprolide acetate] for a period of 3 months prior to surgery, whereas they had not received any hormonal treatment within the 12 months before the surgical procedure.
  Interventions: Drug: Leuprolide Acetate
- GnRH-a - (No Intervention): Group B [GnRHa-] consisted of 30 patients with a mean age of 38 years and a mean BMI of 27 kg/m2. Sixteen of them had stage 2 and 14 had stage 3 endometriosis. They did not receive GnRH-a treatment before operation. In addition, no treatment with oral contraceptives or other therapy was administered within 12 months prior to surgery.

INTERVENTIONS:
Drug: Leuprolide Acetate — Leuprolide acetate was administered 3 months before laparoscopy in women of group A.
  Arms: GnRH-a +

SUMMARY:
Purpose: Neo-angiogenesis is necessary for adhesion and invasiveness of endometriotic lesions in women affected by endometriosis. VEGF is one of the major components of angiogenesis and is part of the major pathway TF-PAR-2-VEGF that leads to neo-angiogenesis. SP1 is a transcriptional factor that has lately been studied for its crucial role in angiogenesis, via a distinct pathway. We hypothesize that by blocking angiogenetic pathways we can repress endometriotic lesions. GnRH-agonists are routinely used, especially pre-operatively, in endometriosis. It would be interesting to clarify which angiogenetic pathways are affected and pave the way for further research over anti-angiogenetic effects on endometriosis.

Methods: We used qRT-PCR to study mRNA expression levels of TF, PAR-2, VEGF and SP1 in endometriotic tissues of women who underwent surgery for endometriosis and received GnRH-a [leuprolide acetate] preoperatively.

DETAILED DESCRIPTION:
The subjects in this study were women of reproductive age. From September 2015 to December 2022, sixty women with known endometriosis [stage 2 and 3], were recruited. Their mean age was 38 years. They were nulliparous and had a mean BMI of 27 kg/m2. The ovarian endometrioma, present in all the participants, was diagnosed by ultrasonography and/or magnetic resonance imaging.

This was a prospective randomized follow up study with analysis of ovarian samples derived from GnRH agonists-treated and non-treated women before surgery. The randomization was performed by accessing a central internet-based randomization program. The random allocation sequence and the assignment of the participants to interventions were made by 2 of the authors [A.K. and S.K].

After enrollment, patients were divided into 2 groups . During laparoscopy, biopsy specimens of the ovarian endometrioma were collected. The staging of endometriosis was based on the rASRM classification system. In group B, surgery was performed during the proliferative phase of the menstrual cycle. All biopsy specimens were collected in accordance with the guidelines of the Declaration of Helsinki and with the approval of the ethical committee of the General University Hospital of Patras. Informed consent was obtained from all women.

ELIGIBILITY:
Inclusion Criteria:

* reproductive age.
* endometriosis [stage 2 and 3]
* nulliparous

Exclusion Criteria:

* women who received any hormonal treatment within the 12 months before the surgical procedure
* obesity BMI>32kg/m2

Ages: 32 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
VEGF | 3 months
  VEGF levels with or without leuprolide acetate treatment
Tissue factor | 3 months
  Tissue factor levels with or without leuprolide acetate treatment
PAR-2 | 3 months
  PAR-2 levels with or without leuprolide acetate treatment
SP1 | 3 months
  SP1 levels with or without leuprolide acetate treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Patras University School of Medicine, Patra, Peloponnese, Greece
- Tottori University Faculty of Medicine, Yonago, Tottori, Japan

IPD SHARING:
Plan to Share IPD: No
Results of this study

REFERENCES:
- [Derived] Filindris T, Papakonstantinou E, Keramida M, Panteris E, Kalogeropoulos S, Georgopoulos N, Taniguchi F, Adonakis G, Harada T, Kaponis A. The effect of GnRH-a on the angiogenesis of endometriosis. Hormones (Athens). 2024 Sep;23(3):509-515. doi: 10.1007/s42000-024-00559-6. Epub 2024 Apr 19. PMID 38639888